CLINICAL TRIAL: NCT06851910
Title: Intravenous Lacosamide for the Treatment of Acute Pain in Trigeminal Neuralgia: A Prospective Observational Study
Brief Title: Intravenous Lacosamide for the Treatment of Acute Pain in Trigeminal Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Albert Muñoz Vendrell, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: EOM043/24
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia; lacosamide; acute treatment; rescue treatment
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Drug: Lacosamide — Patients will be included if they are prescribed intravenous lacosamide for their trigeminal neuralgia exacerbation
  Other Names: Vimpat

SUMMARY:
This prospective observational study evaluates the effectiveness and safety of intravenous lacosamide as a rescue treatment for acute pain in patients presenting to the emergency department with trigeminal neuralgia

DETAILED DESCRIPTION:
This study is a prospective observational investigation evaluating the effectiveness and safety of intravenous lacosamide as a rescue treatment for acute pain exacerbations in trigeminal neuralgia. The trial will be conducted at Hospital Universitari de Bellvitge over a two-year period, enrolling approximately 20 patients who present to the emergency department with acute TN pain and receive intravenous lacosamide based on the treating physician's discretion.

Trigeminal neuralgia is characterized by severe, paroxysmal facial pain, often resistant to conventional therapies. While sodium channel blockers such as carbamazepine and oxcarbazepine are first-line treatments, many patients experience refractory pain or unacceptable side effects. Evidence supporting intravenous options for acute exacerbations remains limited, with studies suggesting potential benefits of phenytoin, lidocaine, and lacosamide. Lacosamide, a voltage-gated sodium channel modulator with a slow inactivation mechanism, has demonstrated efficacy in neuropathic pain and retrospective analyses of TN cases. However, no prospective studies have systematically evaluated its impact in the acute setting.

Data collection will include demographic and clinical variables, TN characteristics, prior treatments, lacosamide infusion parameters, and concurrent medication use. Pain response will be assessed using an 11-point Numerical Pain Rating Scale (NPRS) at baseline, 2 hours post-infusion, at ED discharge, and at 24 hours and 7 days. Additional outcomes include changes in attack frequency, interference with daily activities (Brief Pain Inventory-Facial), patient satisfaction (PGIC), duration of pain relief, and adverse events at multiple time points.

Lacosamide will be administered intravenously per standard clinical practice, with continuous hemodynamic monitoring during and after infusion. Patients will be followed in the ED for at least 2 hours, with structured telephone follow-ups at 24 hours and 7 days post-infusion.

This study aims to generate real-world data on the effectiveness of intravenous lacosamide in acute TN exacerbations. Given the lack of high-quality evidence for emergency pain management in TN, findings may inform future controlled trials and refine clinical recommendations.

ELIGIBILITY:
All patients diagnosed with trigeminal neuralgia who present to the emergency department of Hospital de Bellvitge for an acute pain exacerbation and are prescribed intravenous lacosamide as symptomatic pain treatment, according to the treating physician's discretion, will be considered for inclusion.

Inclusion Criteria:

* Diagnosis of classical or idiopathic trigeminal neuralgia according to the criteria of the International Classification of Headache Disorders (ICHD-3).
* Age over 18 years.
* Signed informed consent.

Exclusion Criteria:

* Contraindication for treatment with lacosamide (previous hypersensitivity reaction, known atrioventricular block).
* Mental or psychiatric illness that interferes with the ability to understand and sign the informed consent.
* Language barrier.
* Lack of cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with primary trigeminal neuralgia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 2 hours post-infusion
  Measured by the Numerical Pain Rating Scale (NPRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). A decrease of ≥50% from baseline indicates improvement in pain intensity.
Adverse effects | Through study completion, an average of 1 week
  Incidence of adverse effects

SECONDARY OUTCOMES:
Sustained pain relief | Through study completion, an average of 1 week
  ≥30%, ≥50% and 75% changes in the numerical pain rating scale (NPRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Reduction in the number of paroxysms.
Impact on daily activities | After 7 days
  Assessed using the Brief Pain Inventory-Facial (BPI-Facial), a 14-question scale measuring pain interference with daily activities. Each question is rated on an 11-point scale from 0 (no interference) to 10 (complete interference), with higher scores indicating greater impairment.
Patient Global Impression of Change | Through study completion, an average of 1 week
  Measured using the 7-point Patient Global Impression of Change (PGIC) scale, which ranges from 1 (very much better) to 7 (very much worse). Lower scores indicate greater perceived improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Muñoz Vendrell, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain